CLINICAL TRIAL: NCT05994534
Title: A Phase 1/2 Pharmacokinetic and Pharmacodynamic Study of NPI-001 Oral Solution Compared to Cysteamine Bitartrate in Cystinosis Patients
Brief Title: PK and PD Study of NPI-001 and Cysteamine Bitartrate
Acronym: INCA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nacuity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-23-01
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cystinosis
MeSH Terms: conditions — Cystinosis | interventions — Cysteamine; N-Acetylcysteinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cysteamine (Active Comparator): Single dose, tablets in current treatment dose
  Interventions: Drug: Cysteamine Bitartrate
- NPI-001 (Experimental): Single dose, NPI-001 (N-acetylcysteine amide) oral solution at molar equivalent of current cysteamine dose.
  Interventions: Drug: N-Acetylcysteine Amide

INTERVENTIONS:
Drug: Cysteamine Bitartrate — Single dose, tablets at current therapeutic dose
  Other Names: Cystagon
  Arms: cysteamine
Drug: N-Acetylcysteine Amide — Single dose, oral solution
  Other Names: NPI-001
  Arms: NPI-001

SUMMARY:
Safety, pharmacokinetics, and pharmacodynamics of NPI-001 oral solution in cystinosis patients compared with cysteamine.

DETAILED DESCRIPTION:
This study will examine the safety, pharmacokinetics, and pharmacodynamics of NPI-001 oral solution in cystinosis patients, aged ≥ 10 years. The ability of NPI-001 to reduce cystine will be assessed and compared with cysteamine.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, any race, ≥ 10 years of age.
2. Diagnosis of nephropathic cystinosis and able to cease cysteamine therapy for 2 days.
3. Females will be nonpregnant and nonlactating, and females of childbearing potential and males will agree to use contraception as detailed in the protocol.
4. Able to comprehend and willing to sign an informed consent /assent form and to abide by the study restrictions (travel as necessary, clinical phase 1 unit or similar for up to 3 days).

Exclusion Criteria:

1. Have undergone kidney transplantation.
2. Are receiving dialysis treatment.
3. History of significant hypersensitivity to NAC or any ingredient of NPI-001 oral solution.
4. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the 30 days prior to Day 1.
5. Inability to provide blood samples, including difficulty with venous access.
6. Subjects who, in the opinion of the Investigator and/or Sponsor (or designee), should not participate in this study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of Cystine Levels Over Time | 1 day
  Cystine concentration over 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hugh McCarthy, PhD, FRACP, Principal Investigator — Sydney Children's Health Network
Locations (1):
- Children's Hospital at Westmead, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.